CLINICAL TRIAL: NCT03663842
Title: Effectiveness of a Novel Neural Tissue Management to Improve Short-term Pain and Disability in Patients With Sciatica
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Principal Investigator, Renato Almeida, Principal Investigator, Centro Universitário Augusto Motta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25/2010
Record Dates: First submitted 2018-09-05; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Sciatica Pain; Physical Therapy Modalities; Manual Therapies; Disability Evaluation
Keywords: Lumbosacral Plexus; Physical Therapy Modalities; Manual Therapies; Disability Evaluation.
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neural tissue management (Experimental): Myofascial release technique; Hip joint mobilization technique; Cross-fiber friction over the sacroiliac joints; Neural mobilization to improve sciatic nerve excursion.
  Interventions: Other: Physical therapy treatment

INTERVENTIONS:
Other: Physical therapy treatment — All patients underwent the same techniques, and there was no modification of the intervention protocol during the study: (1) Myofascial release technique - piriformis muscle and biceps femoral muscle; (2) Hip joint mobilization; (3) Cross-fiber friction over the sacroiliac joints; (4) Neural mobilization to improve sciatic nerve excursion.

SUMMARY:
Objectives: To analyse the effects of sciatic neural mobilisation, in combination to the treatment of the surrounding structures, on pain and disability. Secondly, to investigate baseline characteristics that may be associated with improvements in pain and lumbar disability. Methods: Twenty-eight patients with a clinical diagnosis of sciatica were treated with neural mobilization, joint mobilisation and soft tissue techniques. Pain intensity and lumbar disability were assessed at baseline and after treatment using a Numerical Rating Scale (0-10) and the Oswestry Disability Index (0-100), respectively. The pre- and post-intervention data were compared.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain with radiating leg pain and/or paresthesia below the knee that follows the L5 and/or S1 dermatomal pattern.

Exclusion Criteria:

* History of lumbar and abdominal surgery
* Rheumatologic syndromes (e.g. Rheumatoid arthritis);
* Lumbar stenosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-05-10 (Actual); Primary Completion 2010-11-10 (Actual); Study Completion 2010-12-10 (Actual)

PRIMARY OUTCOMES:
Pain intensity | From enrollment to end of treatment at 12 weeks
  Measured by the Numerical Rating Scale (NRS 0-10)
Lumbar disability | From enrollment to end of treatment at 12 weeks.
  Assessed by the Oswestry Disability Index (ODI).It consists of 10 items addressing different aspects of disability. Each item is scored from 0 to 5, with higher values representing greater disability. The sum of the item scores is divided by the total possible score (50 if all sections are completed), and the resulting total is multiplied by 100 to be described as a percentage score.

CONTACTS AND LOCATIONS:
Overall Officials: Renato Almeida, PhD, Principal Investigator — Centro Universitário Augusto Motta

IPD SHARING:
Plan to Share IPD: No